CLINICAL TRIAL: NCT06985329
Title: Evaluation of Neurocognitive Skills, VisuoSpatial Perception and Perspective Perception in Amputees
Brief Title: 3-Dimensional Evaluation of Body Perception
Status: Not yet recruiting | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu Dilek, Assoc. Prof., Trakya University
Other Study IDs: TÜTFGOBAEK 2025/20
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Body Image; Cognition; Decision Making; Visuospatial/Perceptual Abilities; Neurocognitive Function; Executive Function (Cognition); Amputation
Keywords: Body Image; Cognition; Neuropsychological Test; Amputation; Executive Function; Decision Making; Visuospatial Skills

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amputee Group: Amputees between the ages of 18-65 who use prostheses will be included in the study. Participants who meet the inclusion criteria will be included in this group.
- Control Group: A healthy control group will be recruited. This group will be matched in terms of age, gender, and educational status to the amputee group.

SUMMARY:
The goal of this observational study is to evaluate the changing body perception of amputees aged 18-65 years using prostheses through different personal perspectives of the right-left distinction. In addition, we aimed to examine the relationship between possible changes in body perception and visual spatial perception and neurocognitive performances. The main questions that this study aimed to answer are as follows:

1. Is there a difference between the amputee group and the control group in terms of parameters related to body perception?
2. Is there a difference between the amputee group and the control group in terms of neurocognitive skills?
3. Is there any difference between the amputee group and the control group in terms of visual spatial perception abilities?

To examine whether changes in body perception in amputees affect neurocognitive performance, visuospatial perception and perspective perception and the relationship between them will be compared with a healthy control group.

The assessments to be applied to both groups can be summarised as follows:

* Demographic information such as age, gender, and education level will be recorded.
* Mini-mental state test will be used to assess the cognitive level.
* Edinburgh Handedness Scale will be used to determine the dominant side.
* Right-left discrimination and personal perspective perception will be assessed using a desktop programme.
* The clock drawing test and Benton line orientation test will be used to visual spatial perception.
* A computer based program called The Central Nervous System (CNS) Vital Signs Neurocognitive Test Battery will be used to asesses neurocognitive abilities.

ELIGIBILITY:
Inclusion criteria for the amputee group:

* Acquired amputees
* Aged 18-65 years
* Using a prosthesis for at least six months
* At least a primary school graduate
* Individuals who can adapt to prolonged, attention-demanding activities will be included.
* Standardised Mini Mental State Examination score of >24.

Following the recruitment of the amputee group, a healthy control group will be recruited to match it in terms of age, gender and educational status.

Inclusion criteria for the healthy control group:

* Age range: 18-65 years
* At least a primary school graduate
* Individuals who can adapt to prolonged, attention-demanding activities will be included.
* Standardised Mini Mental State Examination score of >24.

Exclusion criteria for the amputee group:

* Individuals with congenital amputation
* Those with phantom limb pain and/or sensation
* Those with an open wound on the stump
* Bilateral amputation
* Any neurological or psychiatric diagnosis
* Those using sedative medication and/or its derivatives
* Have vision and related problems
* Individuals who are illiterate
* Individuals participating in treatments targeting body representation (e.g. imagery-based treatments or progressive motor visualisation) will not be included in the study.

Exclusion criteria for the Healthy Control Group:

* Having any neurological or psychiatric diagnosis
* Using sedative medication and/or its derivatives
* People with vision and related problems
* Illiterate individuals will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the amputee group, orthotic prosthesis clinics will be contacted in various cities. In order to increase the number of participants, participants will be recruited from other cities outside Edirne. Priority will be given to cities with large populations, such as Istanbul and Ankara.
  Healthy volunteers will be collected within the city of Edirne.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Standardized Mini Mental State Test | 5 minutes
  : It is one of the tests used to assess cognitive impairment. It consists of 5 main topics including various areas of cognitive functioning such as time and space orientation, stored memory, attention and calculation, short-term memory, language (writing sentences, drawing shapes, reading and applying written instructions, etc.). It is aimed to minimize distraction by applying in a quiet environment where the participants are comfortable.
Edinburgh Hand Preference Inventory | 2 minutes
  It is a 10-item scale that assesses participants' dominant hand preference. The researcher directs the items to the participants and the participants are expected to answer "right", "partly right", "left", "partly left" or "I use both".
Clock Drawing Test | 5 minutes
  It is a test that assesses visual-motor functions, planning, sequencing, abstract thinking skills and visual spatial perception. Participants are given a 10 cm hollow circle on paper. Participants are asked to place all the numbers of the clock inside the circle and draw the hour and minute hands so that the hour and minute hands point to 10 minutes past 11.
Benton Line Orientation Test | 15-20 minutes
  It is a test used to measure the orientation component of visual spatial abilities. It consists of 5 practice tests and 30 test items. Participants who get at least 2 of the 5 practice tests correct will be directed to move on to the 30 test items. In this test, participants are asked to: Perceive which 2 lines in the lower part of the test item are in equal angle and direction with which two of the 11 lines in the upper part of the test item and mark the 2 numbers with the correct option.
CNS Vital Signs Test | 25 minutes
  It is a computer-based neurocognitive test battery used to assess participants' neurocognitive performance. It consists of 7 sub-headings in total and evaluates 12 neurocognitive domains of the participants. The 7 sub-headings are as follows; verbal memory, visual memory, finger tapping, symbol-number coding, stroop test, attention orientation, continuous performance tests. The tests are conducted on a computer. The participant is expected to complete the tests by following the rules and instructions specified in each test.
Evaluation of Perspective Perception | 10-15 minutes
  A virtual reality supported desktop application developed with a software program will be used to evaluate perspective perception. Participants are asked to stand in front of the computer positioned on the desktop. During the test, the participants will see an avatar animation in different angles (0-45-90-135-180-225-270-315) and perspectives (eye level, above eye level, below eye level, from the top and from the bottom) and they will be asked to adapt the body of the avatar they see to their own body and make the same limb movement (shoulder abduction) that the avatar makes. At the end of the test, movement angle values and reaction times of the participants will be recorded.
Right-left Discrimination Test | 5-10 minutes
  As an alternative to Recognise, the paradigm developed with the "e-prime" software program will be used to evaluate the right-left distinction. Participants will be presented with hand visuals with mental rotation categorized from easy to difficult. Test categories will be applied in a randomized order. In each set (easy-moderate-difficult), 30 images will be presented in different postures and randomly right and left. The participants will answer the presented images by pressing the "right" or "left" buttons on the screen. Participants will be asked to complete the test as soon as they can. At the end of the test, participants' completion times, reaction times for each level and side, and success rates will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rosen AB, McGrath ML, Maerlender AL. Males with chronic ankle instability demonstrate deficits in neurocognitive function compared to control and copers. Res Sports Med. 2021 Mar-Apr;29(2):116-128. doi: 10.1080/15438627.2020.1723099. Epub 2020 Jan 29. PMID 31992081
- [Background] Gualtieri CT, Johnson LG. Reliability and validity of a computerized neurocognitive test battery, CNS Vital Signs. Arch Clin Neuropsychol. 2006 Oct;21(7):623-43. doi: 10.1016/j.acn.2006.05.007. Epub 2006 Oct 2. PMID 17014981
- [Background] Dilek B, Tavli EY, Yilmaz E, Yaşar E, Ocal T, Çetinkaya O, et al. A Mobile Application Program that Configures Right-Left Hand Recognition According to the Degree of Mental Rotation Difficulty. 2024 Medical Technologies Congress (TIPTEKNO). 2024. IEEE. p.1-3. doi:
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Molloy DW, Alemayehu E, Roberts R. Reliability of a Standardized Mini-Mental State Examination compared with the traditional Mini-Mental State Examination. Am J Psychiatry. 1991 Jan;148(1):102-5. doi: 10.1176/ajp.148.1.102. PMID 1984692
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204